CLINICAL TRIAL: NCT03864939
Title: Randomized Pilot Study to Improve Postprostatectomy Incontinence and Potency by Application of Dried Human Amnion Graft
Brief Title: Application of Dried Human Amnion Graft to Improve Postprostatectomy Incontinence and Potency
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: German Centre for Assessment and Evaluation of Innovative Techniques in Medicine (Other)
Responsible Party: Principal Investigator, Dimitri Barski, Principal Investigator, Lukas-Krankenhaus GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAM01
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Continence; Potency; Complication; Biochemical Recurrence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are blinded during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dHAM (Experimental): dHAM wrap is placed during RRP.
  Interventions: Drug: dHAM
- Standard (Placebo Comparator): A standard RRP is performed.
  Interventions: Drug: No dHAM

INTERVENTIONS:
Drug: dHAM — A dehydrated human amnion membrane (dHAM, 1x3cm) is placed around the neurovascular bundle (NVB) on the left and right side and vesicourethral anastomosis (VUA) during radical retropubic prostatectomy (RRP).
  Arms: dHAM
Drug: No dHAM — A standard radical retropubic prostatectomy (RRP) without dHAM is performed (Walsh, 2005).
  Arms: Standard

SUMMARY:
The investigators present a randomized trial of patients undergoing placement of dehydrated human amnion membrane (dHAM) around the neurovascular bundle (NVB) and vesicourethral anastomosis (VUA) during radical retropubic prostatectomy (RRP) in a tertiary center in Germany.

DETAILED DESCRIPTION:
Patients suffer under incontinence and impotence after RRP, improving techniques and studies are missing. The human amniotic membrane includes growth factors and unique immune tolerance which can improve tissue regeneration. The preliminary studies could prove the potential value of dHAM in the reconstruction of the urinary tract and nerve protection. The investigators initially present a randomized trial to improve postoperative continence and potency of patients undergoing placement of dehydrated human amnion membrane (dHAM) around the neurovascular bundle (NVB) and vesicourethral anastomosis (VUA) during RRP for the treatment of prostate cancer. RRP is performed in a standardized way by one experienced surgeon. The patients are randomized 1:1 to dHAM vs. placebo and blinded during the study period. The primary outcome is a postoperative continence measure as 24hrs pad test up to 12mos postoperatively. Secondary outcomes are potency, insufficiency of VUA, postoperative complications and biochemical recurrence. Using the T-test with an alpha of 0.05 and a power of 80% and expecting a drop-out of 20% of the patients, an adjusted sample size per arm of 164 patients is required.

ELIGIBILITY:
Inclusion Criteria:

* patients with localized prostate cancer
* indication for radical prostatectomy
* no other treatment of prostate cancer
* availability to informed consent

Exclusion Criteria:

* preoperative incontinence (24hrs pad-test)
* preoperative erectile dysfunction (IIEF-5 < 20)
* metastasized or locally advanced prostate cancer in preoperative assessment
* previous radiation of pelvis
* previous prostate cancer therapy
* psychiatric disease
* participation at another study

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in urine loss | From baseline (1 week after surgery) to 3 weeks after surgery
  Urine loss is assessed by 24 hrs pad-test (in gram)
Change in urine loss | From baseline (1 week after surgery) to 6 weeks after surgery
  Urine loss is assessed by 24 hrs pad-test (in gram)
Change in urine loss | From baseline (1 week after surgery) to 3 months after surgery
  Urine loss is assessed by 24 hrs pad-test (in gram)
Change in urine loss | From baseline (1 week after surgery) to 12 months after surgery
  Urine loss is assessed by 24 hrs pad-test (in gram)

SECONDARY OUTCOMES:
Change in erectile function (EF) | From baseline (4 weeks before surgery) to 6 weeks after surgery
  EF is assessed by IIEF-5 (the International Index of Erectile Function) questionnaire.
Change in erectile function (EF) | From baseline (4 weeks before surgery) to 3 months after surgery
  EF is assessed by IIEF-5 (the International Index of Erectile Function) questionnaire.
Change in erectile function (EF) | From baseline (4 weeks before surgery) to 12 months after surgery
  EF is assessed by IIEF-5 (the International Index of Erectile Function) questionnaire.
Postoperative catheter removal | through study completion, an average of 1 year
  Time of postoperative catheter removal (days)
Complications | perioperative, at 6 weeks, 3 months and 12 months
  Complications are assessed according to Clavien-Dindo classification.
Biochemical recurrence | at 6 weeks, 3 months and 12 months
  Measurement of prostate-specific antigen (PSA)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Barski, PhD, Principal Investigator — Department of Urology, Lukas Hospital Neuss
Locations (1):
- Department of Urology, Lukas Hospital, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Andersson KE, Apostolidis A, Birder L, Bliss D, Brubaker L, Cardozo L, Castro-Diaz D, O'Connell PR, Cottenden A, Cotterill N, de Ridder D, Dmochowski R, Dumoulin C, Fader M, Fry C, Goldman H, Hanno P, Homma Y, Khullar V, Maher C, Milsom I, Newman D, Nijman RJM, Rademakers K, Robinson D, Rosier P, Rovner E, Salvatore S, Takeda M, Wagg A, Wagner T, Wein A; members of the committees. 6th International Consultation on Incontinence. Recommendations of the International Scientific Committee: EVALUATION AND TREATMENT OF URINARY INCONTINENCE, PELVIC ORGAN PROLAPSE AND FAECAL INCONTINENCE. Neurourol Urodyn. 2018 Sep;37(7):2271-2272. doi: 10.1002/nau.23551. Epub 2018 Aug 14. No abstract available. PMID 30106223
- [Background] Asimakopoulos AD, Miano R, Galfano A, Bocciardi AM, Vespasiani G, Spera E, Gaston R. Retzius-sparing robot-assisted laparoscopic radical prostatectomy: Critical appraisal of the anatomic landmarks for a complete intrafascial approach. Clin Anat. 2015 Oct;28(7):896-902. doi: 10.1002/ca.22576. Epub 2015 Jul 21. PMID 26194970
- [Background] Barski D, Gerullis H, Ecke T, Varga G, Boros M, Pintelon I, Timmermans JP, Otto T. Human Amniotic Membrane Is Not Suitable for the Grafting of Colon Lesions and Prevention of Adhesions in a Xenograft Rat Model. Surg Innov. 2017 Aug;24(4):313-320. doi: 10.1177/1553350617709828. Epub 2017 May 26. PMID 28548553
- [Background] Barski D, Gerullis H, Ecke T, Varga G, Boros M, Pintelon I, Timmermans JP, Otto T. Human amniotic membrane dressing for the treatment of an infected wound due to an entero-cutaneous fistula: Case report. Int J Surg Case Rep. 2018;51:11-13. doi: 10.1016/j.ijscr.2018.08.015. Epub 2018 Aug 13. PMID 30130666
- [Background] Barski D, Gerullis H, Ecke T, Varga G, Boros M, Pintelon I, Timmermans JP, Winter A, Bagner JW, Otto T. Repair of a vesico-vaginal fistula with amniotic membrane - Step 1 of the IDEAL recommendations of surgical innovation. Cent European J Urol. 2015;68(4):459-61. doi: 10.5173/ceju.2015.683. Epub 2015 Nov 13. PMID 26855802
- [Background] Barski D, Gerullis H, Ecke T, Yang J, Varga G, Boros M, Pintelon I, Timmermans JP, Otto T. Bladder Reconstruction with Human Amniotic Membrane in a Xenograft Rat Model: A Preclinical Study. Int J Med Sci. 2017 Mar 11;14(4):310-318. doi: 10.7150/ijms.18127. eCollection 2017. PMID 28553162
- [Background] Capogrosso P, Salonia A, Briganti A, Montorsi F. Postprostatectomy Erectile Dysfunction: A Review. World J Mens Health. 2016 Aug;34(2):73-88. doi: 10.5534/wjmh.2016.34.2.73. Epub 2016 Aug 23. PMID 27574591
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Lemke A, Ferguson J, Gross K, Penzenstadler C, Bradl M, Mayer RL, Gerner C, Redl H, Wolbank S. Transplantation of human amnion prevents recurring adhesions and ameliorates fibrosis in a rat model of sciatic nerve scarring. Acta Biomater. 2018 Jan 15;66:335-349. doi: 10.1016/j.actbio.2017.11.042. Epub 2017 Nov 28. PMID 29191510
- [Background] Ogaya-Pinies G, Kadakia Y, Palayapalayam-Ganapathi H, Woodlief T, Jenson C, Syed J, Patel V. Use of Scaffolding Tissue Biografts To Bolster Vesicourethral Anastomosis During Salvage Robot-assisted Prostatectomy Reduces Leak Rates and Catheter Times. Eur Urol. 2018 Jul;74(1):92-98. doi: 10.1016/j.eururo.2016.10.004. Epub 2016 Oct 14. PMID 27751731
- [Background] Ogaya-Pinies G, Palayapalam-Ganapathi H, Rogers T, Hernandez-Cardona E, Rocco B, Coelho RF, Jenson C, Patel VR. Can dehydrated human amnion/chorion membrane accelerate the return to potency after a nerve-sparing robotic-assisted radical prostatectomy? Propensity score-matched analysis. J Robot Surg. 2018 Jun;12(2):235-243. doi: 10.1007/s11701-017-0719-8. Epub 2017 Jun 27. PMID 28656504
- [Background] Patel VR, Samavedi S, Bates AS, Kumar A, Coelho R, Rocco B, Palmer K. Dehydrated Human Amnion/Chorion Membrane Allograft Nerve Wrap Around the Prostatic Neurovascular Bundle Accelerates Early Return to Continence and Potency Following Robot-assisted Radical Prostatectomy: Propensity Score-matched Analysis. Eur Urol. 2015 Jun;67(6):977-980. doi: 10.1016/j.eururo.2015.01.012. Epub 2015 Jan 19. PMID 25613153
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Walsh PC. Re: Anatomical radical retropubic prostatectomy: detailed description of the surgical technique. J Urol. 2005 Jan;173(1):324. doi: 10.1097/01.ju.0000148246.73337.ad. No abstract available. PMID 15592108
- [Derived] Barski D, Gerullis H, Ecke T, Boros M, Brune J, Beutner U, Tsaur I, Ramon A, Otto T. Application of Dried Human Amnion Graft to Improve Post-Prostatectomy Incontinence and Potency: A Randomized Exploration Study Protocol. Adv Ther. 2020 Jan;37(1):592-602. doi: 10.1007/s12325-019-01158-3. Epub 2019 Nov 28. PMID 31782131
- See also: Abrams P, Cardozo L, Khoury S, Wein A. 2005. Incontinence Basics& Evaluation, 3rd International Consultation on Incontinence. Chapter 13: Imaging and other Investigations. — https://www.ics.org/Publications/ICI_3/v1.pdf/chap13.pdf